CLINICAL TRIAL: NCT04358445
Title: Effects of Magnesium-rich Artificial Cerebrospinal Fluid on the Incidence of Cerebral Vasospasm and Clinical Prognosis of Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Application of Magnesium-rich Artificial Cerebrospinal Fluid in Aneurysmal Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJYFY-2019N28
Record Dates: First submitted 2020-03-16; First posted 2020-04-24 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-03

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Non randomized， non parallelized and history case-controled quasi-experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historical control group (No Intervention): The patients were treated by aneurysm clipping in our hospital in the previous nine months, and normal saline (0.9% Sodium Chloride Injection) had applied as intraoperative perfusion solution in operation of the historical control group. All of the 35 patients selected should meet the inclusion and exclusion criteria of this study.
- MACSF group (Experimental): Use Magnesium-Rich Artificial Cerebrospinal Fluid (MACSF) in the operation, and the remaining treatments should strictly follow the guidelines as same as the historical control group.
  Interventions: Other: Magnesium-Rich Artificial Cerebrospinal Fluid

INTERVENTIONS:
Other: Magnesium-Rich Artificial Cerebrospinal Fluid — The Magnesium-Rich Artificial Cerebrospinal Fluid (MACSF) is composed of several qualified clinical intravenous injections according to a specific formula, which has similar physical and chemical properties to physiological CSF. MACSF will be freshly made and used. It will be prepared by trained professionals on a specific workbench and sent to the operating room in a special container. Finally, it will be used in the operation by the neurosurgeons. Aseptic principles should be enforced strictly during the whole procedures, including preparation, transportation and application.
  Arms: MACSF group

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) is a common type of acute hemorrhagic stroke. One of its complications, cerebral vasospasm (CVS), is the main cause of death and disability, with an incidence of up to 30%-90%. Blood and its metabolites are vital reasons for CVS. Normal saline, as an intraoperative irrigation fluid for the surgery of aneurysm clipping, can induce secondary damage to the brain. In this study, a new type of magnesium-rich artificial cerebrospinal fluid (MACSF) has been designed, which has similar ionic concentration, pH value and osmotic pressure compared with the physiological cerebrospinal fluid. It has been confirmed by animal experiments that MACSF can relieve the hyper-responsiveness of cerebral arteries to ET and 5-HT induced by hemorrhagic CSF from patients with aSAH by down-regulating the expression of ETA, contractile ETB and 5-HT1B receptors in the previous research. Therefore, MACSF may have potential effects on preventing and treating CVS. In this study, we plan to apply MACSF as an intraoperative irrigation fluid for the surgery of aneurysm clipping (MACSF group), which is compared with normal saline (historical control group). To evaluate the effects of MACSF on reducing the incidence of CVS and improving the clinical prognosis of patients with aSAH, the occurrence of CVS within 14 days after aneurysm clipping, NIHSS score, as well as mRS scores at 1, 3 and 6 months after aSAH will be recorded and compared. CVS related biomarkers will be used to evaluate the relationship between the occurrence of CVS and the levels of biomarkers in both CSF and blood samples from MACSF group.

DETAILED DESCRIPTION:
From now on, participants who meet the inclusion and exclusion criteria in our hospital will be recruited in the intervention group, if they and their relatives are willing to join in the study. For the historical control group, in which patients were treated by aneurysm clipping in Department of Neurosurgery of the First Affiliated Hospital of Xi'an Jiaotong University during the previous nine months, normal saline (0.9% Sodium Chloride Injection) was applied as intraoperative perfusion solution for their operation. For the intervention group, MACSF will be used. (The composition and concentration of MACSF is as follows: Na+: 146.2 mEq/l, K+: 2.7 mEq/l, Mg2+: 4.2 mEq/l, Cl-: 123 mEq/l, HCO3-: 23.2 mEq/l, Glucose: 0.75 g/l. MACSF is prepared by the staff of Pharmacy Intravenous Admixture Services of First Affiliated Hospital of Xi'an Jiaotong University, according to a specific formula in the specific working area. The whole procedure follow the aseptic principles strictly. Fresh-made MACSF will be placed in a specific container and send to the operating room through specific channels.) Then, for the patients who have signed the informed consent, blood (6ml) and CSF (3ml) samples will be collected during and every other day after the surgery for 14 days. The blood samples should be drawn into a non-anticoagulant tube and a heparin anticoagulant tube respectively. All the samples will be transferred to BioBank of the First Affiliated Hospital of Xi'an Jiaotong University in a liquid nitrogen tank. After re-melted in a water bath of 37℃, the CSF and blood samples will be centrifuged at 4℃ for 10min at 2000r/min, and then the supernatant will be collected and stored at -80℃. At the end of this study, the contents of NPY，MMP-9，MIF，TNF-α，Mg2+ and Ca2+in the samples will be detected by ELISA or mass spectrometry. Transcranial Doppler (TCD) will be observed within 14 days after the operation (daily for the first three days and every other day for the following days). CVS will be diagnosed by TCD, the diagnostic criteria will be described later. CT scan of the brain should be done at least once a week and rechecked anytime when necessary. If there is new low-density lesions, delayed cerebral infarction (DCI) will be diagnosed. The prognosis will be assessed at 1, 3 and 6 months after aSAH onset according to modified Rankin Scale (mRS) . Meanwhile, some indicators will be used to evaluate the safety of MACSF application, which incluiding secondary infection, fluctuation of intracranial pressure and hypermagnesemia. The diagnostic criteria and the solutions will be described in the next part.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 80 years of old;
* aSAH is diagnosed by CTA, DSA or other cranial imaging examination;
* Patient is admitted to hospital within 72 hours after aSAH onset;
* Aneurysm is clipped within 36 hours after admission;
* Patient and his/her relatives are informed and agree to accept the above treatment plan.

Exclusion Criteria:

* Cause of the SAH is not rupture of an intracranial aneurysm;
* Time from SAH onset to admission is longer than 72 hours;
* Time from admission to surgery is longer than 36 hours;
* The patient dose not choose clipping;
* Patient has other serious diseases, such as heart failure, kidney failure, liver failure, etc;
* Patient or his/her relatives refuse to accept the above research plan.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of CVS during and after operation | Within 14 days after surgery
  Transcranial Doppler (TCD) will be used to evaluate the occurrence and severity of CVS, which will be diagnosed according to the following criteria for TCD. First, the mean blood flow velocity of tested arteries is higher than 120cm/s. Second, the mean blood flow velocity of tested arteries increases more than 15cm/s or 20% compared with the previous time. Third, the Lindeggard Index (mean blood flow velocity of MCA/mean blood flow velocity of ipsilateral eICA) is higher than 3
mRS (modified Rankin Scale） | Day 30
  Assess patients' prognosis by the score of modified Rankin Scale.In the mRS, the lowest score is 0, and the highest score is 5. A score of 0 indicates the patients have no symptoms at all, and a score of 5 indicates the patients have severe disability, bed rest, incontinence, and need for continuous care and attention. In this study, we evaluate patient's outcomes by the following criteria. Favorable outcome was defined as mRS<3, whereas poor outcome was mRS≥3.
mRS (modified Rankin Scale） | Day 60
  Assess patients' prognosis by the score of modified Rankin Scale.In the mRS, the lowest score is 0, and the highest score is 5. A score of 0 indicates the patients have no symptoms at all, and a score of 5 indicates the patients have severe disability, bed rest, incontinence, and need for continuous care and attention. In this study, we evaluate patient's outcomes by the following criteria. Favorable outcome was defined as mRS<3, whereas poor outcome was mRS≥3.
mRS (modified Rankin Scale） | Day 90
  Assess patients' prognosis by the score of modified Rankin Scale.In the mRS, the lowest score is 0, and the highest score is 5. A score of 0 indicates the patients have no symptoms at all, and a score of 5 indicates the patients have severe disability, bed rest, incontinence, and need for continuous care and attention. In this study, we evaluate patient's outcomes by the following criteria. Favorable outcome was defined as mRS<3, whereas poor outcome was mRS≥3.

SECONDARY OUTCOMES:
Levels of biomarkers in cerebrospinal fluid (CSF) | Within 14 days after surgery
  Cerebrospinal fluid samples were collected during and every other day after surgery for 14 days to evaluated the effect of MACSF on Neuropeptide Y (NPY, ng/L), Matrix Metalloproteinase-9(MMP-9, ng/L), Macrophage Migration Inhibitory Factor (MIF, ng/L), Tumor Necrosis Factor-α(TNF-α, ng/L).
Levels of ion concentration in cerebrospinal fluid (CSF) | Within 14 days after surgery
  Cerebrospinal fluid samples were collected during and every other day after surgery for 14 days to evaluated the effect of MACSF on Mg2+ (mEq/L)and Ca2+ (mEq/L).
Levels of biomarkers in blood | Within 14 days after surgery
  Blood samples were collected during and every other day after surgery for 14 days to evaluated the effect of MACSF on Neuropeptide Y (NPY, ng/L), Matrix Metalloproteinase-9(MMP-9, ng/L), Macrophage Migration Inhibitory Factor (MIF, ng/L), Tumor Necrosis Factor-α(TNF-α, ng/L).
Levels of ion concentration in blood | Within 14 days after surgery
  Blood samples were collected during and every other day after surgery for 14 days to evaluated the effect of MACSF on Mg2+ (mEq/L)and Ca2+ (mEq/L).
Duration of hospitalization | up to 60 days
  Length of hospital stay in the intensive care unit, total length of hospital stay, the days of anti-CVS drugs use, etc

OTHER OUTCOMES:
Incidence and severity of MACSF-induced infection | up to 14 days
  If the patient has some symptoms of infection, the doctor in charge must determine whether it is MACSF-induced infection and assess the severity. First, the MACSF-induced infection will be diagnosed by the patient's symptoms and the MACSF sample's pathogenic detection. Second, the severity of infection will be evaluated by the indicators including the duration of fever, the kinds of antibiotics, the duration of antibiotics use and the results of CSF examination
Fluctuation of intracranial pressure（ICP） | up to 14 days
  ICP will be assessed by invasive ICP monitoring and lumbar puncture. The severity will be evaluated by days of use of dehydrated drugs
Incidence of hypermagnesemia | up to 14 days
  Pay close attention to the clinical manifestations of fatigue, disappearance of tendon reflex and decreased blood pressure, and monitor the blood electrolyte level dynamically to assess the incidence of hypermagnesemia

CONTACTS AND LOCATIONS:
Overall Officials: Luo Guogang, MD,PHD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Cheng Y, Han X, Xie W, Xu G, Bai X, Qi L, Zhang L, Liu R, Dong W, Feng W, Pang C, Zhang W, Liu F, Cao X, Xu Y, Luo G. Safety and efficacy of magnesium-rich artificial cerebrospinal fluid for subarachnoid hemorrhage. Front Neurol. 2024 Mar 28;15:1376216. doi: 10.3389/fneur.2024.1376216. eCollection 2024. PMID 38606277